CLINICAL TRIAL: NCT00110617
Title: A Randomized, Open-label, Multi-center, Phase II Study to Evaluate the Safety and Efficacy of Deferasirox (ICL670) 20 mg/kg/Day Relative to Subcutaneous Deferoxamine in Sickle Cell Disease Patients With Iron Overload From Repeated Blood Transfusions
Brief Title: Study of Deferasirox Relative to Subcutaneous Deferoxamine in Sickle Cell Disease Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: External Affairs, Novartis Pharmaceuticals
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CICL670A2201
Record Dates: First submitted 2005-05-10; First posted 2005-05-11 (Estimated); Results first posted 2011-05-02 (Estimated); Last update posted 2011-05-26 (Estimated); Status verified 2011-05

CONDITIONS: Sickle Cell Disease; Iron Overload; Hemolytic Anemia
Keywords: Sickle Cell Disease; Iron Overload from Repeated Blood Transfusions; Iron Overload; Blood Transfusions
MeSH Terms: conditions — Anemia, Sickle Cell; Iron Overload; Anemia, Hemolytic | interventions — Deferasirox; Deferoxamine

ARMS (2):
- Deferasirox (ICL670) (Experimental): Deferasirox (ICL670) 20 mg/kg orally once daily for 104 weeks.
  Interventions: Drug: Deferasirox (ICL670)
- Deferoxamine (DFO) then ICL670 (Experimental): Deferoxamine (DFO) subcutaneously for a weekly dose of 175 mg/kg for 24 weeks then crossed over to receive Deferasirox (ICL670) orally 20 mg/kg for a total of 104 weeks on therapy.
  Interventions: Drug: Deferasirox (ICL670); Drug: Deferoxamine (DFO)

INTERVENTIONS:
Drug: Deferasirox (ICL670) — Deferasirox was provided in 125 mg, 250 mg, and 500 mg dispersible tablets and was administered orally at an initial dose of 20 mg/kg/day.
Drug: Deferoxamine (DFO) — Deferoxamine was supplied in vials of 500 mg and 2000 mg administered subcutaneously for a weekly dose of 175 mg/kg.
  Arms: Deferoxamine (DFO) then ICL670

SUMMARY:
This study will examine the long-term safety and efficacy of Deferasirox in patients with sickle cell disease and iron overload from repeated blood transfusions.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 2 years
* Male or female patients with sickle cell disease (SS, SC, SD, Sβo or Sβ+ thalassemia)
* Iron overload from repeated blood transfusion, as defined by one of the following:

  1. For patients > 16 years old receiving simple transfusions: lifetime history of receipt of at least 120 ml/kg or 30 adult units of packed red blood cells, OR
  2. For patients ≤ 16 years old receiving simple transfusions: lifetime history of receipt of at least 120 ml/kg of packed red blood cells, OR
  3. For all patients receiving exchange transfusions in the absence of a previous attempt to achieve negative iron balance: lifetime performance of at least 20 procedures, OR
  4. For all patients: liver iron content ≥ 7 mg Fe/g dry weight as measured by biopsy, Magnetic Resonance Imaging (MRI), or magnetic susceptibility performed within 3 months prior to entry into screening
* For entry into the screening period: serum ferritin of ≥ 1000 µg/mL on at least two occasions during the prior year obtained in the absence of concomitant infection.
* Body weight > 10 kg
* No known allergy or contraindication to the administration of deferoxamine
* Ability to comply with all study-related procedures, medications, and evaluations
* Sexually active pre-menopausal female patients must use double-barrier contraception, oral contraceptive plus barrier contraceptive, or must have undergone clinically documented total hysterectomy and/or oophorectomy, tubal ligation or be postmenopausal defined by amenorrhea for at least 12 months.
* Written informed consent by the patient or for pediatric patient's consent of the patient's legal guardian. The definition of the term 'pediatric' for enrollment and study conduct will be in accordance with the local legislation.

Exclusion Criteria:

* Serum creatinine above the upper limit of normal
* Significant proteinuria
* History of nephrotic syndrome
* Alanine aminotransferase (ALT) ≥ 250 U/L at screening
* Clinical evidence of active hepatitis B or hepatitis C
* History of HIV
* Fever or other signs/symptoms of infection within 10 days prior to the screening visit
* Uncontrolled systemic hypertension
* History of Myocardial Infarction, Congestive Heart Failure or unstable cardiac disease not controlled by standard medical therapy
* Clinically relevant cataract or a previous history of clinically relevant ocular toxicity related to iron chelation
* Presence of a surgical or medical condition that might significantly alter the absorption, distribution, metabolism or excretion of any study drug
* History of drug or alcohol abuse within the 12 months prior to enrollment
* Pregnant or breast feeding patients
* Patients treated with systemic investigational drug within 4 weeks prior or with topical investigational drug 7 days prior to the screening visit
* Randomization in a previous clinical trial involving ICL670

Other protocol-related inclusion / exclusion criteria may apply.

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 212 (Actual)
Dates: Start 2005-05; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (59):
- United States (56):
  - University of Alabama Pediatric Hematology/Oncology, Birmingham, Alabama
  - University of Alabama Medical center, Birmingham, Alabama
  - University of South Alabama Medical Center, Mobile, Alabama
  - University of South Alabama, Mobile, Alabama
  - Loma Linda University Medical Center, Loma Linda, California
  - Children's Hospital Oakland, Oakland, California
  - Center for Cancer and Blood Disorders, Washington D.C., District of Columbia
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Howard University Hospital, Washington D.C., District of Columbia
  - Miami Children's Hospital, Miami, Florida
  - Tampa Children's Hospital at St Joseph's, Tampa, Florida
  - Tampa Children's Hospital at St. Joseph's, Tampa, Florida
  - H. Lee Muffit Cancer Center and Research Institute/James A. Haley Veterans Hospital, Tampa, Florida
  - Emory University School of Medicine, Atlanta, Georgia
  - Children's Healthcare of Atlanta at Scottish Rite, Atlanta, Georgia
  - Adult Sickle Cell Clinic, Augusta, Georgia
  - Backus Children's Hospital, Savannah, Georgia
  - University of Illinois at Chicago, Chicago, Illinois
  - Children's Memorial Hospital, Chicago, Illinois
  - Pediatric Sickle Cell Program/James Whitcomb Riley Hospital for Children, Indianapolis, Indiana
  - St. Jude Children's Hospital Affiliate, Baton Rouge, Louisiana
  - Tulane University Sickle Cell Center, New Orleans, Louisiana
  - Children's Hospital, New Orleans, Louisiana
  - LSU Health Sciences Center/Carroll W. Feist Professor of Cancer Research, Shreveport, Louisiana
  - Brigham and Woman's Hospital/Harvard Medical School, Boston, Massachusetts
  - Children's Hospital Boston, Boston, Massachusetts
  - Children's Hospital, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Karmanos Cancer Institute, Detroit, Michigan
  - Washington University School of Medicine, St Louis, Missouri
  - SUNY Downstate Medical Center, Brooklyn, New York
  - New York Methodist Hospital, Brooklyn, New York
  - Weill Medical College of Cornell University, New York, New York
  - Columbia University, New York, New York
  - Sickle Cell Center, Montefiore Hospital, The Bronx, New York
  - Carolinas Medical Transplant Center, Charlotte, North Carolina
  - University of Cincinnati, Cincinnati, Ohio
  - Children's Hospital Medical Center, Cincinnati, Ohio
  - The University of Oklahoma, Oklahoma City, Oklahoma
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Pennsylvania Oncology/Hematology, Philadelphia, Pennsylvania
  - Jefferson University, Philadelphia, Pennsylvania
  - Drexel University College of Medicine, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Hillman Cancer Center, Pittsburgh, Pennsylvania
  - Liberty Hematology Oncology Center, Columbia, South Carolina
  - Palmetto Health Clinical Trials, Columbia, South Carolina
  - Santee Hematology/Oncology, Sumter, South Carolina
  - St Jude's Children's Research Hospital, Memphis, Tennessee
  - St. Jude's Children Research Hospital, Memphis, Tennessee
  - Cooks Children's Hospital, Fort Worth, Texas
  - Texas Children's Hospital/Baylor College of Medicine, Houston, Texas
  - Scott and White Memorial Hospital & Clinics, Temple, Texas
  - Children's Hospital of the King's Daughter, Norfolk, Virginia
  - Medical College of Virginia, Richmond, Virginia
  - Virginia Commonwealth University, Richmond, Virginia
- Canada (3):
  - University of Alberta, Edmonton, Alberta
  - The Ottawa Hospital, Ottawa, Ontario
  - Hopital Ste-Justine, Montreal, Quebec

REFERENCES:
- See also: Visit NovartisClinicalTrials.com: Pre-qualify for a trial, and view a list of trials and participating study centers. — http://www.novartisclinicaltrials.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 212 participants were enrolled in the study; however, 9 participants from Site 512 were excluded due to severe Good Clinical Practice (GCP) violations. 203 participants are included in the Full Analysis Set 1.
Period: Overall Study
Arm/Group | Deferasirox (ICL670) | Deferoxamine (DFO) Then ICL670
Started | 135 | 68 (Full Analysis Set 1 does not include 9 participants who were excluded due to GCP violations.)
Safety Set 1; Received Study Drug | 135 | 56
Full Analysis 2; Received ICL670 | 135 | 53
On Going at Week 24 | 126 | 53
Completed | 96 | 39
Not Completed | 39 | 29
Not completed — Adverse Event | 2 | 4
Not completed — Abnormal Laboratory Value | 4 | 2
Not completed — Lack of Efficacy | 1 | 0
Not completed — Patient no longer requires study drug | 1 | 0
Not completed — Protocol Violation | 5 | 0
Not completed — Withdrawal by Subject | 10 | 4
Not completed — Lost to Follow-up | 9 | 1
Not completed — Administrative problems | 6 | 5
Not completed — Death | 1 | 1
Not completed — Did not receive study drug | 0 | 12

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Deferasirox (ICL670) | Deferoxamine (DFO) Then ICL670 | Total
Number analyzed (Participants) | 135 | 68 | 203
Age Continuous [Mean (Standard Deviation); unit: years] | 16.4 (10.31) | 16.2 (10.15) | 16.3 (10.23)
Age, Customized [Number; unit: participants]
  2- < 6 Years | 6 | 4 | 10
  6- <12 Years | 42 | 21 | 63
  12- <16 Years | 35 | 18 | 53
  16- < 50 Years | 50 | 24 | 74
  50- <65 Years | 2 | 1 | 3
  = 65 Years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 56 | 33 | 89
  Male | 79 | 35 | 114
Race/Ethnicity, Customized [Number; unit: Participants]
  Caucasian | 2 | 0 | 2
  Black | 130 | 65 | 195
  Oriental | 0 | 0 | 0
  Other | 3 | 3 | 6
Weight Group [Number; unit: Participants]
  <15 kg | 0 | 0 | 0
  15- <35 kg | 39 | 23 | 62
  35- < 55 kg | 43 | 18 | 61
  55- <75 kg | 42 | 22 | 64
  =75 kg | 10 | 3 | 13
  Missing | 1 | 2 | 3

OUTCOME MEASURES:

1. Secondary Outcome: Absolute Change in Serum Ferritin From Baseline to Week 24
Description: Absolute change from baseline serum ferritin after 24 weeks of treatment with Deferasirox (ICL670) and absolute change from baseline serum ferritin after 24 weeks of treatment with Deferoxamine. Means were adjusted for the amount of transfused blood.
Time Frame: Baseline, 24 Weeks
Population: Per protocol- 1 defined as all participants who had study drug and had an assessment of serum ferritin at Baseline and at Week 24.
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/mL
Arm/Group | Deferasirox (ICL670) | Deferoxamine (DFO) Then ICL670
Number analyzed (Participants) | 117 | 50
mg/mL | -173.2 [-691.5 to 345.1] | -868.7 [-1661.9 to 75.5]

2. Secondary Outcome: Absolute Change in Serum Ferritin After Start of Treatment With Deferasirox (ICL670) to Week 24 and to Week 52
Description: Absolute change in serum ferritin after start of treatment with Deferasirox (ICL670) to week 24 and the absolute change in serum ferritin after start of treatment with Deferasirox (ICL670) to week 52 for the Deferasirox treatment group and the Deferoxamine then Deferasirox treatment group. Means were adjusted for the amount of transfused blood.
Time Frame: Start of Deferasirox (ICL670) treatment, 24 Weeks, 52 Weeks
Population: Per Protocol- 2 set defined as all participants who received study drug and had an assessment of serum ferritin at Start of ICL670 treatment and at 24 weeks or 52 weeks.
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/mL
Arm/Group | Deferasirox (ICL670) | Deferoxamine (DFO) Then ICL670
Number analyzed (Participants) | 113 | 49
mg/mL
  24 weeks from ICL670 treatment start (n=111,47) | -146.7 [-673.7 to 380.2] | -204.7 [-1014.7 to 605.3]
  52 weeks from ICL670 treatment start (n=113,40) | -487.3 [-761.6 to -213.0] | -545.7 [-1007.1 to -84.2]

3. Primary Outcome: The Number of Participants With Adverse Events (AEs) in the First 24 Weeks of Treatment
Description: The number of participants with Adverse Events (AEs) overall and according to Medical Dictionary for Regulatory Activities (MedDRA) preferred term greater than or equal to 5% participants in any group by treatment in the first 24 weeks.
Time Frame: 24 Weeks
Population: Safety-1 set: All participants, except participants enrolled in Center 512, who received at least one dose of study medication during the first 24 weeks.
Measure: Number; unit: participants
Arm/Group | Deferasirox (ICL670) | Deferoxamine (DFO) Then ICL670
Number analyzed (Participants) | 135 | 56
participants
  Headache | 30 | 17
  Sickle cell anaemia with crisis | 30 | 8
  Diarrhoea | 30 | 5
  Vomiting | 21 | 9
  Pyrexia | 19 | 9
  Nausea | 20 | 4
  Abdominal pain | 16 | 6
  Upper respiratory tract infection | 10 | 9
  Rash | 14 | 3
  Cough | 10 | 7
  Constipation | 11 | 2
  Pain in Extremity | 10 | 3
  Back Pain | 8 | 4
  Chest Pain | 7 | 5
  Oropharyngeal pain | 7 | 5
  Pruritus | 7 | 5
  Abdominal pain upper | 8 | 3
  Nasal congestion | 6 | 4
  Urinary tract infection | 9 | 0
  Arthralgia | 7 | 1
  Nasopharyngitis | 4 | 3
  Insomnia | 3 | 3
  Dizziness | 2 | 3
  Injection site pain | 0 | 3

4. Secondary Outcome: Absolute Change in Serum Ferritin After Start of Treatment With Deferasirox (ICL670) to Week 104
Description: Absolute change in serum ferritin after start of treatment with Deferasirox (ICL670) to week 104 for the Deferasirox treatment group. Means were adjusted for the amount of transfused blood.
Time Frame: Start of Deferasirox (ICL670) treatment, 104 Weeks
Population: Per Protocol- 2 set defined as all participants who received study drug and had assessment of serum ferritin at Start of ICL670 treatment and at 104 weeks.
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/mL
Arm/Group | Deferasirox (ICL670)
Number analyzed (Participants) | 87
mg/mL | -682.6 [-1090.3 to -274.9]

ADVERSE EVENTS:
Groups:
- Period 1 Deferasirox (ICL670): Period 1 (first 24 weeks) Deferasirox (ICL670) 20 mg/kg orally once daily.
- Period 1 Deferoxamine (DFO): Period 1 (first 24 weeks) Deferoxamine (DFO) subcutaneously for a weekly dose of 175 mg/kg.
- Period 2 Deferasirox (ICL670): Period 2 (after 24 weeks) Deferasirox (ICL670) 20 mg/kg orally once daily.
- Period 2 Deferoxamine (DFO) Then ICL670: Period 2 (After 24 weeks) DFO group cross over to Deferasirox (ICL670) orally 20 mg/kg completing 52 weeks on therapy and then entering an extension period.
Arm/Group | Period 1 Deferasirox (ICL670) | Period 1 Deferoxamine (DFO) | Period 2 Deferasirox (ICL670) | Period 2 Deferoxamine (DFO) Then ICL670
Serious Adverse Events (participants affected / at risk) | 40/135 | 20/56 | 78/135 | 22/53
Other Adverse Events (participants affected / at risk) | 91/135 | 39/56 | 118/135 | 44/53
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Period 1 Deferasirox (ICL670) (N=135) | Period 1 Deferoxamine (DFO) (N=56) | Period 2 Deferasirox (ICL670) (N=135) | Period 2 Deferoxamine (DFO) Then ICL670 (N=53)
Acute chest syndrome (Blood and lymphatic system disorders) | 0 | 2 | 2 | 1
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0 | 3 | 1
Cardio-respiratory arrest (Cardiac disorders) | 1 | 0 | 1 | 1
Conduction disorder (Cardiac disorders) | 0 | 0 | 0 | 1
Intracardiac thrombus (Cardiac disorders) | 0 | 0 | 0 | 1
Sickle cell anaemia (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 1
Sickle cell anaemia with crisis (Congenital, familial and genetic disorders) | 27 | 6 | 38 | 11
Adrenocortical insufficiency acute (Endocrine disorders) | 0 | 0 | 0 | 1
Photophobia (Eye disorders) | 0 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 0 | 6 | 1
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 2 | 1
Inguinal hernia (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 5 | 0 | 6 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 4 | 0 | 7 | 1
Asthenia (General disorders) | 0 | 1 | 0 | 0
Catheter site pain (General disorders) | 0 | 1 | 1 | 0
Chest pain (General disorders) | 1 | 0 | 7 | 4
Chills (General disorders) | 0 | 1 | 0 | 1
Device breakage (General disorders) | 0 | 0 | 0 | 1
Device malfunction (General disorders) | 0 | 1 | 0 | 1
Implant site reaction (General disorders) | 0 | 1 | 0 | 0
Oedema peripheral (General disorders) | 1 | 0 | 2 | 0
Pain (General disorders) | 2 | 0 | 3 | 1
Pyrexia (General disorders) | 6 | 3 | 17 | 6
Cholelithiasis (Hepatobiliary disorders) | 0 | 1 | 3 | 1
Bacteraemia (Infections and infestations) | 0 | 0 | 0 | 2
Bacterial infection (Infections and infestations) | 1 | 0 | 1 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 2 | 0
Catheter site infection (Infections and infestations) | 0 | 1 | 0 | 1
Cellulitis (Infections and infestations) | 0 | 2 | 0 | 0
Device related infection (Infections and infestations) | 1 | 0 | 3 | 0
Gastroenteritis (Infections and infestations) | 1 | 0 | 3 | 1
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 1 | 0
Infected skin ulcer (Infections and infestations) | 0 | 0 | 1 | 0
Lobar pneumonia (Infections and infestations) | 1 | 0 | 1 | 0
Mycoplasma infection (Infections and infestations) | 0 | 0 | 1 | 0
Parvovirus infection (Infections and infestations) | 0 | 0 | 1 | 0
Pharyngitis (Infections and infestations) | 0 | 0 | 3 | 0
Pharyngitis streptococcal (Infections and infestations) | 1 | 1 | 2 | 0
Pneumonia (Infections and infestations) | 4 | 0 | 9 | 4
Pneumonia klebsiella (Infections and infestations) | 1 | 0 | 1 | 0
Pneumonia streptococcal (Infections and infestations) | 0 | 0 | 1 | 0
Pyelonephritis (Infections and infestations) | 0 | 0 | 0 | 1
Rotavirus infection (Infections and infestations) | 0 | 0 | 1 | 0
Sepsis (Infections and infestations) | 0 | 0 | 2 | 0
Septic shock (Infections and infestations) | 1 | 0 | 1 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 1 | 0
Staphylococcal bacteraemia (Infections and infestations) | 0 | 0 | 1 | 1
Streptococcal infection (Infections and infestations) | 0 | 0 | 1 | 0
Tooth abscess (Infections and infestations) | 0 | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 2 | 4 | 1
Urinary tract infection (Infections and infestations) | 2 | 0 | 4 | 1
Viral infection (Infections and infestations) | 1 | 1 | 2 | 0
Clavicle fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0
Fibula fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Patella fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 1 | 1 | 1 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 2 | 0
Blood culture positive (Investigations) | 2 | 0 | 2 | 0
Blood pressure diastolic decreased (Investigations) | 1 | 0 | 1 | 0
Culture throat positive (Investigations) | 1 | 0 | 2 | 0
Haemoglobin decreased (Investigations) | 0 | 1 | 1 | 0
Heart rate increased (Investigations) | 1 | 0 | 1 | 0
Hepatic enzyme increased (Investigations) | 2 | 0 | 2 | 0
Liver function test abnormal (Investigations) | 2 | 0 | 2 | 0
Oxygen saturation decreased (Investigations) | 0 | 0 | 1 | 1
Serum ferritin increased (Investigations) | 0 | 0 | 1 | 0
Urine protein/creatinine ratio increased (Investigations) | 0 | 0 | 1 | 0
White blood cells urine positive (Investigations) | 1 | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0
Haemosiderosis (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hyperglycaemic hyperosmolar nonketotic syndrome (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0
Arthropathy (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 2 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1 | 0
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 0 | 5 | 0
Altered state of consciousness (Nervous system disorders) | 1 | 0 | 1 | 0
Ataxia (Nervous system disorders) | 0 | 0 | 1 | 0
Balance disorder (Nervous system disorders) | 0 | 0 | 1 | 0
Carotid artery occlusion (Nervous system disorders) | 0 | 0 | 1 | 0
Cerebral ischaemia (Nervous system disorders) | 0 | 1 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 1 | 1
Convulsion (Nervous system disorders) | 1 | 0 | 4 | 0
Dysarthria (Nervous system disorders) | 0 | 0 | 2 | 0
Headache (Nervous system disorders) | 2 | 2 | 5 | 1
Hypokinesia (Nervous system disorders) | 0 | 0 | 1 | 0
Loss of consciousness (Nervous system disorders) | 0 | 0 | 1 | 0
Migraine (Nervous system disorders) | 2 | 0 | 2 | 0
Moyamoya disease (Nervous system disorders) | 1 | 0 | 1 | 0
Nervous system disorder (Nervous system disorders) | 0 | 0 | 0 | 1
Syncope (Nervous system disorders) | 0 | 0 | 1 | 1
Transient ischaemic attack (Nervous system disorders) | 2 | 0 | 2 | 1
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 1
Confusional state (Psychiatric disorders) | 0 | 0 | 1 | 0
Delirium (Psychiatric disorders) | 1 | 0 | 1 | 0
Mental status changes (Psychiatric disorders) | 0 | 0 | 1 | 0
Haematuria (Renal and urinary disorders) | 1 | 0 | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 1 | 0
Renal failure acute (Renal and urinary disorders) | 0 | 0 | 1 | 0
Renal papillary necrosis (Renal and urinary disorders) | 0 | 0 | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 3 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 3 | 0
Pharyngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 2
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Poor peripheral circulation (Vascular disorders) | 0 | 0 | 0 | 1
Superior vena caval occlusion (Vascular disorders) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Period 1 Deferasirox (ICL670) (N=135) | Period 1 Deferoxamine (DFO) (N=56) | Period 2 Deferasirox (ICL670) (N=135) | Period 2 Deferoxamine (DFO) Then ICL670 (N=53)
Sickle cell anaemia with crisis (Congenital, familial and genetic disorders) | 7 | 4 | 17 | 7
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 4 | 4
Abdominal pain (Gastrointestinal disorders) | 14 | 6 | 30 | 8
Abdominal pain upper (Gastrointestinal disorders) | 7 | 3 | 13 | 5
Constipation (Gastrointestinal disorders) | 11 | 2 | 24 | 4
Diarrhoea (Gastrointestinal disorders) | 30 | 5 | 36 | 9
Nausea (Gastrointestinal disorders) | 16 | 4 | 33 | 10
Vomiting (Gastrointestinal disorders) | 18 | 9 | 30 | 11
Chest pain (General disorders) | 6 | 5 | 16 | 9
Injection site pain (General disorders) | 0 | 3 | 0 | 0
Oedema peripheral (General disorders) | 0 | 0 | 7 | 1
Pain (General disorders) | 0 | 0 | 11 | 1
Pyrexia (General disorders) | 14 | 7 | 34 | 15
Hypersensitivity (Immune system disorders) | 0 | 0 | 7 | 3
Gastroenteritis (Infections and infestations) | 0 | 0 | 1 | 4
Influenza (Infections and infestations) | 0 | 0 | 4 | 3
Nasopharyngitis (Infections and infestations) | 4 | 3 | 18 | 6
Otitis media (Infections and infestations) | 0 | 0 | 4 | 3
Pharyngitis streptococcal (Infections and infestations) | 0 | 0 | 6 | 5
Pneumonia (Infections and infestations) | 0 | 0 | 2 | 4
Sinusitis (Infections and infestations) | 0 | 0 | 9 | 2
Upper respiratory tract infection (Infections and infestations) | 10 | 7 | 25 | 7
Urinary tract infection (Infections and infestations) | 7 | 0 | 17 | 6
Transfusion reaction (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 3
Alanine aminotransferase increased (Investigations) | 0 | 0 | 7 | 1
Blood pressure diastolic increased (Investigations) | 0 | 0 | 8 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 7 | 1 | 20 | 5
Back pain (Musculoskeletal and connective tissue disorders) | 7 | 3 | 20 | 11
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 9 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 10 | 3 | 31 | 9
Dizziness (Nervous system disorders) | 2 | 3 | 8 | 0
Headache (Nervous system disorders) | 28 | 15 | 47 | 13
Insomnia (Psychiatric disorders) | 3 | 3 | 7 | 1
Dysuria (Renal and urinary disorders) | 0 | 0 | 7 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 10 | 7 | 29 | 14
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 7 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 8 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 6 | 4 | 20 | 7
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 6 | 5 | 24 | 5
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 9 | 2
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 3 | 3
Pruritus (Skin and subcutaneous tissue disorders) | 7 | 5 | 13 | 2
Rash (Skin and subcutaneous tissue disorders) | 14 | 3 | 21 | 4

LIMITATIONS AND CAVEATS:
Due to severe good clinical practice violations, data from 9 participants recruited for Center 512 was excluded from the main analysis of the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.